CLINICAL TRIAL: NCT04880681
Title: Evaluation of Length and Quality of Prostate Biopsies Taken by a New Biopsy Needle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: double needle
Record Dates: First submitted 2021-05-05; First posted 2021-05-11 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer (Diagnosis)
Keywords: Prostatic Neoplasms; Neoplasms; Genital Neoplasms, Male; Urogenital Neoplasms; Neoplasms by Site; Prostatic Diseases
MeSH Terms: conditions — Prostatic Neoplasms; Disease; Neoplasms; Genital Neoplasms, Male; Urogenital Neoplasms; Neoplasms by Site; Prostatic Diseases | interventions — Biopsy, Needle

STUDY DESIGN:
Intervention Model Description: 60 patients eligible for prostate biopsy are randomized into 2 arms (30+30 patients) using either the novel needle and actuator device or standard Tru Cut needle and actuator device used in the clinic today. On average 12 biopsies are taken from each patient. Biopsy length (primary outcome) is evaluated by a pathologist who is blinded to device used.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient and pathologist are unaware of which needle/device is used. All biopsies are taken from behind the back of the patient enabling masking from the patient. To assess masking success, patients will be asked to guess which device was used after the procedure is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novel needle (Experimental): Novel needle (18 G, 25 cm with 19 mm sample notch) in a new actuator.
  Interventions: Device: Novel needle (18 G, 25 cm with 19 mm sample notch) in a new actuator.
- Standard Tru Cut needle (Active Comparator): Standard tru cut biopsy needle (Argon 18G, 25 cm biopsy needle with a 19 mm sample notch) in a standard actuator (Möller Medical Blue RBG-1000-10-1000).
  Interventions: Device: Standard Tru Cut biopsy needle (Argon 18G, 25 cm biopsy needle with a 19 mm sample notch) in a standard actuator (Möller Medical Blue RBG-1000-10-1000)

INTERVENTIONS:
Device: Novel needle (18 G, 25 cm with 19 mm sample notch) in a new actuator. — Trans Rectal Ultrasound guided Prostate Biopsy using the assigned needle. Approximately 12 biopsies per patient.
  Other Names: prostate biopsy
  Arms: Novel needle
Device: Standard Tru Cut biopsy needle (Argon 18G, 25 cm biopsy needle with a 19 mm sample notch) in a standard actuator (Möller Medical Blue RBG-1000-10-1000) — Trans Rectal Ultrasound guided Prostate Biopsy using the assigned needle. Approximately 12 biopsies per patient.
  Other Names: prostate biopsy
  Arms: Standard Tru Cut needle

SUMMARY:
Patient-blinded randomized controlled trial evaluating length and quality of prostate biopsies taken by a novel biopsy needle.

DETAILED DESCRIPTION:
Prostate biopsy is the golden standard for prostate cancer diagnosis. Transrectal prostate biopsy (TRUSbx) is the most widely used technique. The biopsy chamber of the Tru Cut needle is in general 19 mm. However, it is on average filled only with 13 mm of tissue. Biopsy length is strongly correlated with diagnostic accuracy of prostate cancer.

Additionally, TRUSbx has a high risk of infection due to bacteria being brought across the colon wall. The investigators have shown that a new needle design reduces this bacterial transfer in an ex vivo setting and a previous trial (NCT049091230) has shown non inferior biopsy length when compared to the standard Tru Cut needle. A further improvement of the needle has now been designed aiming to increase biopsy length and quality, with the possible potential to improve prostate cancer diagnosis. This is the first human pilot aiming to evaluate if biopsy length of the novel needle is superior to a standard Tru Cut biopsy needle in prostate biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for prostate biopsy
* Signed informed written consent

Exclusion Criteria:

- None (other than general contraindications for prostate biopsy or patient not willing to participate)

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Prostate biopsy length (measured by pathologist) | within 21 days post biopsy
  Length of biopsy specimen in millimeters

SECONDARY OUTCOMES:
Prostate biopsy fragmentation | within 21 days post biopsy
  The number of sections the biopsy specimen is made of
General appearance of biopsy assessed by pathologist (biopsy quality) | within 21 days post biopsy
  General quality of biopsy specimen on a scale from 0-3 (no biopsy, poor, good, excellent)
Prostate biopsy length (measured in biopsy needle chamber) | within 21 days post biopsy
  Length of biopsy specimen in millimeters
Prostate biopsy length (measured after removal from biopsy chamber) | within 21 days post biopsy
  Length of biopsy specimen in millimeters

OTHER OUTCOMES:
Pain from biopsy sampling | At the time of biopsy sampling
  Numeric rating Pain Scale rating from 0-10
14 day complications | 14 days after biopsy
  Any complications related to the biopsy (example infection, bleeding)
30 day complications | 30 days after biopsy
  Any complications related to the biopsy (example infection, bleeding)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Linder, Ass prof, Principal Investigator — Lund University
Locations (1):
- Helsingborg Hospital, Helsingborg, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Forsvall A, Fisher J, Wagenius M, Broman C, Korkocic D, Bratt O, Linder A. Prostate biopsy quality and patient experience with the novel Forsvall biopsy needle - a randomized controlled non-inferiority trial. Scand J Urol. 2021 Jun;55(3):235-241. doi: 10.1080/21681805.2021.1921024. Epub 2021 May 17. PMID 33999764
- [Result] Forsvall A, Fisher J, Cardoso JFP, Wagenius M, Tverring J, Nilson B, Dahlin A, Bratt O, Linder A, Mohanty T. Evaluation of the Forsvall biopsy needle in an ex vivo model of transrectal prostate biopsy - a novel needle design with the objective to reduce the risk of post-biopsy infection. Scand J Urol. 2021 Jun;55(3):227-234. doi: 10.1080/21681805.2021.1921023. Epub 2021 May 17. PMID 33999753
- See also: Forsvall et al. Prostate biopsy quality and patient experience with the novel Forsvall biopsy needle - a randomized controlled non-inferiority trial. — https://pubmed.ncbi.nlm.nih.gov/33999764/
- See also: Forsvall et al, Evaluation of the Forsvall biopsy needle in an ex vivo model of transrectal prostate biopsy — https://pubmed.ncbi.nlm.nih.gov/33999753/